CLINICAL TRIAL: NCT05054543
Title: A Phase 3 Randomized, Double-Blinded Bridging Trial to Evaluate the Efficacy of Uproleselan Administered With Chemotherapy Versus Chemotherapy Alone in Chinese Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Study to Evaluate the Efficacy of Uproleselan in Combination With Chemotherapy in Chinese Patients With R/R AML
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In light of the strategic realignment of the company's development focus, it has been determined to discontinue the further development of Uproleselan Injection.
Sponsor: Apollomics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APL-106-02
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory AML
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — uproleselan; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uproleselan (Experimental): Uproleselan in combination with mitoxantrone, etoposide and cytarabine (MEC) during induction; Uproleselan in combination with HiDAC/IDAC during consolidation
  Interventions: Drug: Uproleselan
- Placebo (Saline, 0.9% Sodium Chloride) (Placebo Comparator): Placebo in combination with mitoxantrone, etoposide and cytarabine (MEC) during induction; Placebo in combination with HiDAC/IDAC during consolidation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Uproleselan — A rationally designed E-selectin antagonist used to inhibit binding of cells to E-selectin
  Other Names: GMI-1271
  Arms: Uproleselan
Drug: Placebo — 0.9% Sodium Chloride
  Other Names: Saline
  Arms: Placebo (Saline, 0.9% Sodium Chloride)

SUMMARY:
This bridging study will evaluate the efficacy of uproleselan, a specific E-selectin antagonist, in combination with chemotherapy to treat Chinese relapsed/refractory AML patients, compared to chemotherapy alone. The safety of uproleselan when given with chemotherapy will also be investigated in patients with relapsed/refractory AML

DETAILED DESCRIPTION:
This trial will enroll approximately 140 randomized subjects 18 through 75 years of age at the time of randomization with primary refractory AML or relapsed AML (first or second untreated relapse) and eligible to receive induction chemotherapy as described.

Randomization will be done at trial entry at a 1:1 ratio, and will be stratified by age (<60, ≥60 years) and disease status (primary refractory/early relapse ≤6 months, late relapse>6 months) and prior HSCT status. Treatment assignment received at randomization will be maintained during all induction and consolidation cycles.

This trial will have the following sequential phases: screening, baseline, induction treatment and count recovery, response assessment, consolidation treatment (if remission is achieved), and follow-up for relapse and survival assessment. Subjects not achieving remission will continue to be followed for long-term trial endpoints such as disease progression and survival. Blinding will be maintained until database lock. This study will carry out long-term follow-up for all subjects for a maximum of 3 years or death of subjects or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years and ≤75 years in age
2. AML diagnosed with ≥20% myeloid marrow blasts or peripheral blood blasts per WHO criteria(2008) at the time of initial diagnosis
3. For subjects with primary refractory AML:

   1. Refractory disease is defined as persistent disease (≥5% blasts in the bone marrow) at least 28 days after initiation of anthracycline-containing induction therapy or relapse from a first remission (CR, CRi, complete remission with incomplete platelet recovery [CRp], CRh) lasting for <90 days. Isolated extramedullary disease is not allowed.
   2. Persistent disease (≥5% blasts in the bone marrow): Must have received 1 (and only 1) prior anthracycline-containing induction regimen. Except as defined below, a second induction with intent to induce remission is not allowed.

      1. Re-induction within 28 days with a comparable regimen containing the same chemotherapy agents (e.g., cytarabine/daunorubicin '7+3' and '5+2'; or cytarabine/daunorubicin '7+3' and '7+3') is allowed.
      2. Re-induction within 28 days with a comparable regimen using an alternative anthracycline (e.g., cytarabine/daunorubicin in the first induction and cytarabine/idarubicin in the second) is allowed.
      3. Previous induction with certain regimens (venetoclax/hypomethylating agent [HMA], venetoclax/LDAC, single agent HMA) followed by an anthracycline induction regimen is allowed. May have achieved remission with certain regimens (venetoclax/HMA, venetoclax/LDAC, single agent HMA) and then experience relapse now refractory to anthracycline-containing induction.
   3. Relapse from first remission (CR, CRi, CRp, CRh) lasting <90 days: 1) After achieving first remission from any induction regimen, may have received consolidation before experiencing relapse.
4. No more than one prior stem cell transplant.
5. Has not received the chemotherapy regimen to be used for induction on this trial.
6. Is considered medically eligible to receive the chemotherapy regimen to be used for induction on this trial.
7. Peripheral absolute blast count (ABC) ≤40.0 x 109/L (ABC = total white blood cells [WBC] x blast % in peripheral blood). Hydroxyurea to control absolute blast count is allowed prior to uproleselan/placebo dosing.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia
2. Acute leukemia of ambiguous lineage (biphenotypic leukemia)
3. Chronic myeloid leukemia with myeloid blast crisis
4. Active signs or symptoms of CNS involvement by malignancy (No lumbar puncture required)
5. Prior use of G-CSF, CM-CSF or plerixafor within 7 days of dosing.
6. Allogeneic HSCT ≤ 4 months, autologous HSCT ≤ 3 months or donor lymphocyte infusion (DLI) ≤ 6 weeks prior to Uproleselan/placebo dosing.
7. Any immunotherapy or radiotherapy therapy within 28 days of dosing; any other experimental therapy or chemotherapy within 14 days of dosing
8. Inadequate organ function.
9. Abnormal liver function.
10. Known active infection with hepatitis A, B, or C, or human immunodeficiency virus.
11. Creatinine clearance <45 mL/min (Cockcroft-Gault method) or creatinine >1.5x ULN (any assessed must be within eligibility limit).
12. Uncontrolled acute life-threatening bacterial, viral, or fungal infection.
13. Myocardial infarction within 6 months of uproleselan/placebo dosing, or subject has current significant cardiovascular disease.
14. Major surgery within 4 weeks before uproleselan/placebo dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Time from the date of randomization into the study to the date of death.

SECONDARY OUTCOMES:
Remission rate(rate of CR, CR/CRi and CR/CRh) | Up to 60 days
  Defined as the rate of subjects who reach CR, CR/CRi and CR/CRh
Duration of remission | Up to 3 years
  Time from date of first documented remission to date of relapse or death from any cause, whichever occurs first.
Event-free survival | Up to 3 years
  Time from date of randomization into the study to the date of treatment failure, relapse, or death from any cause; whichever occurs first.
Rate of severe oral mucositis | Up to 254 days
  Incidence of severe oral mucositis experienced in patients after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, PhD, Principal Investigator — Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University, Hangzhou

IPD SHARING:
Plan to Share IPD: No